CLINICAL TRIAL: NCT01336959
Title: A Two-part, Randomized, Double-blind, Placebo-controlled, Single Dose Study of BCT197 for the Prevention of Acute Kidney Injury (AKI) in Patients Undergoing Elective Cardiac Surgery With Cardiopulmonary Bypass (CPB)
Brief Title: Safety & Efficacy of BCT197 in Patients Undergoing Cardiac Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBCT197A2202; 2011-002735-25 (EudraCT Number)
Record Dates: First submitted 2011-04-13; First posted 2011-04-18 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Cardiopulmonary Bypass; CABG; Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open Label - BCT197 Part A (Experimental): 10mg single dose of BCT197
  Interventions: Drug: BCT197 Part A
- BCT197 Part B (Experimental): Single dose of 50mg BCT197
  Interventions: Drug: BCT197 Part B
- BCT 197 Placebo Part B (Placebo Comparator): Single dose of matching placebo to 50mg BCT197
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCT197 Part A — open label single dose administration of 10mg BCT197, 2 hours prior to surgery
  Arms: Open Label - BCT197 Part A
Drug: Placebo — Single dose matching placebo administered 2 prior to surgery
  Arms: BCT 197 Placebo Part B
Drug: BCT197 Part B — BCT197 50mg single dose administered 2 hours prior to surgery
  Arms: BCT197 Part B

SUMMARY:
This study will assess the safety and efficacy of BCT197 on acute kidney injury in patients undergoing cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cardiac surgery with CPB. Allowable procedures are CABG alone, aortic valve replacement or repair alone, mitral valve replacement or repair alone, CABG with aortic valve replacement or repair, and CABG with mitral valve replacement or repair. Patients with repeat surgery for any of the procedures can be included.
* Patients must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) 18 kg/m2
* Have an eGFR ≥ 30 and ≤ 60 mL/min/1.73 m2 to participate in Part A, or an eGFR > 60 mL/min/1.73 m2 to participate in Part B. Upon completion of Part A, patients with eGFR ≥ 30 mL/min/1.73 m2 may participate in Part B, with dose administered as per the dosing table

Exclusion Criteria:

* left ventricular ejection fraction, in the last 6 months, ≥30%
* Active systemic infection or uncontrolled diabetes mellitus with a glucose ≥250 mg% at the screening assessment
* Pregnant or nursing (lactating) women,
* Female subjects must either:

have been surgically sterilized or hysterectomized at least 6 months prior to study participation, or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to study participation. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow- up hormone level assessment is she considered not of child bearing potential, Surgical sterilization procedures or hysterectomy must be supported with clinical documentation made available to the sponsor and noted in the Relevant Medical History / Current Medical Conditions section of the CRF, OR be postmenopausal. Female subjects are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms). Female subjects 60 years of age or younger must confirm menopause by the demonstration of a plasma FSH level in the postmenopausal range according to the lab normal range. Documentation of a prior plasma FSH level is acceptable

* History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of drug abuse as indicated by the laboratory assays conducted during screening or baseline
* New cancer diagnosis with planned chemotherapy and/or radiation therapy, or cancer requiring ongoing chemotherapy and/or radiation therapy at the time of screening

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Parkin, PhD FRCP, Study Director — Mereo BioPharma
Locations (13):
- United States (6):
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Wynnewood, Pennsylvania
  - Novartis Investigative Site, Falls Church, Virginia
- Israel (6):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Herzliya
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BCT197 Part A: 10 mg BCT197 dosed 2 hours prior to surgery
- BCT197 Part B: BCT197 Part B: Randomized Double-blind BCT197. Single dose 50mg capsule given 2 hours prior to surgery
- Placebo Part B: Double-blind randomized Placebo: Placebo capsules matching 50mg BCT197 capsules. Single dose given 2 hours prior to surgery
Period: Overall Study
Arm/Group | BCT197 Part A | BCT197 Part B | Placebo Part B
Started | 8 | 42 | 41
Completed | 8 | 37 | 40
Not Completed | 0 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Open Label - BCT197: BCT197 Part A
- Randomized Double-blind BCT197: BCT197 Part B: Randomized Double-blind BCT197
- Randomized Double-blind BCT 197 Placebo: Placebo: Placebo capsules
- Total: Total of all reporting groups
Arm/Group | Open Label - BCT197 | Randomized Double-blind BCT197 | Randomized Double-blind BCT 197 Placebo | Total
Number analyzed (Participants) | 8 | 42 | 41 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 26 | 27 | 57
  >=65 years | 4 | 16 | 14 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 10 | 25
  Male | 2 | 33 | 31 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 41 | 40 | 89
  Black | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Renal Function Measured at 48 Hours Post Cardiac Surgery With Cardiopulmonary Bypass Pump.
Description: Median percent change from baseline in estimated Glomerular Filtration Rate (eGFR) at 48 hours postdose.
Time Frame: 48 hours
Population: Full Analysis Set
Measure: Median (5% Confidence Interval); unit: Median percentage change
Arm/Group | Open Label - BCT197 | Randomized Double-blind BCT197 | Randomized Double-blind BCT 197 Placebo
Number analyzed (Participants) | 8 | 42 | 41
Median percentage change | 8.68 [-45.2 to 30.06] | 77 [32.52 to 142.36] | 85.81 [55.08 to 132.44]

2. Secondary Outcome: Pharmacokinetic Measurements of Drug in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass Pump. Pharmacokinetics Will be Measured Using Cmax
Description: Max serum concentration reached (ng/mL)
Time Frame: 4 days
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BCT197 Part A | BCT197 Part B | Placebo Part B
Number analyzed (Participants) | 8 | 32 | 0
ng/mL | 64.5 (33.1) | 206 (64.4) |

ADVERSE EVENTS:
Arm/Group | Open Label - BCT197 | Randomized Double-blind BCT197 | Randomized Double-blind BCT 197 Placebo
Serious Adverse Events (participants affected / at risk) | 1/8 | 13/42 | 7/41
Other Adverse Events (participants affected / at risk) | 0/8 | 37/42 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label - BCT197 (N=8) | Randomized Double-blind BCT197 (N=42) | Randomized Double-blind BCT 197 Placebo (N=41)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Enterobacter test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label - BCT197 (N=8) | Randomized Double-blind BCT197 (N=42) | Randomized Double-blind BCT 197 Placebo (N=41)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 16 (16) | 11 (11)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 11 (11) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 5 (5) | 6 (6)
Generalised oedema (General disorders) | 0 (0) | 6 (6) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 5 (5)
Pain (General disorders) | 0 (0) | 3 (3) | 3 (3)
Secretion discharge (General disorders) | 0 (0) | 2 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 6 (6) | 7 (7)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (3)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 8 (8) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 7 (7) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 2 (2)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 7 (7) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 9 (9) | 4 (4)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (2) | 5 (5)
Breath sounds abnormal (Investigations) | 0 (0) | 5 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Calcium ionised decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 6 (6) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)
Labile blood pressure (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)
Pallor (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Polyuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
The trial was terminated early after a planned interim analysis due to the lack of benefit of BCT197 in preventing acute kidney injury.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs must seek written permission from the sponsor prior to publication on any trial results.